CLINICAL TRIAL: NCT02962934
Title: An Observational Pharmacokinetic Sudy of Ceftolozane-Tazobactam in Intensive Care Unit in Patients With and Without Continuous Renal Replacement Therapy.
Brief Title: An Observational Pharmacokinetic Sudy of Ceftolozane-Tazobactam in Intensive Care Unit in Patients With and Without CRRT
Acronym: CT-PK
Status: Completed | Type: Observational
Sponsor: Royal Brisbane and Women's Hospital (Other Government)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Jason Roberts, Professor, Royal Brisbane and Women's Hospital
Other Study IDs: Royal_Brisbane
Record Dates: First submitted 2016-11-01; First posted 2016-11-15 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Gram-Negative Bacterial Infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, blood and ultrafiltrate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non CRRT group: Critically ill patients receiving Ceftolozane-Tazobactam not receiving continuous renal replacement therapy
  Interventions: Other: Non CRRT group
- CRRT group: Critically ill patients receiving Ceftolozane-Tazobactam who require continuous renal replacement therapy
  Interventions: Other: CRRT group

INTERVENTIONS:
Other: Non CRRT group — Non CRRT group:Blood samples prior to first dose of Ceftolozane-Tazobactam and at 15, 45, 1hr, 2hr 3hr 4h 5h 6h 7h 8h.
  Groups: Non CRRT group
Other: CRRT group — CRRT group: Pre and Post dialysis filter blood samples taken prior to first dose of Ceftolozane-tazobactam and at 15min, 45min, 1h 2h 3h 4h 5h 6h 7h 8h.
  Ultrafiltrate samples at 1 hr,2h 4h 6h 8h
  Groups: CRRT group

SUMMARY:
The purpose of this study is to try to find out how critically ill patients receiving the antibiotic, ceftolozane-tazobactam, process it in their body. Investigators would like to study if the antibiotic concentrations during a dose of this antibiotic reaches the right concentrations necessary to kill the bacteria that is causing the infection. The process by which a drug travels through the body in blood, how it is broken down and removed by the body is called pharmacokinetics (PK). We can measure the PK by taking blood samples at specific times after the antibiotic is given.

Investigators would like to do the study in patients receiving dialysis and patients who are not receiving dialysis. This information about how the antibiotic is processed in the critically ill patient is unknown and it is important to know whether the doses doctors give patients to fight infection are adequate. If antibiotic concentrations are low in the blood, it gives the bacteria an opportunity to become resistant to the antibiotic which can lead to the antibiotic being less effective against bacteria potentially exposing future patients with infections to a limited range of effective antibiotics.

Patients will be consented, and given the antibiotic as prescribed. Blood samples will be taken from the drip that is already in the patients arm just as the antibiotic starts, at 15 and 45 minutes, at 1,2,3,4,5,6,7 and 8 hours. Patients who are on dialysis will have the blood samples taken from the dialysis machine before the blood reaches the dialysis filter (same blood samples as the non dialysis patients) and also bloods samples taken after the filter at 45 minutes, 2 and 6 hours. Dialysis patients will also have 5 separate samples of ultrafiltrate taken (approximately 10mls) - ultrafiltrate is the waste product of the dialysis process. The total amount of blood will be 40mls which is equal to about 2 tablespoons. The dialysis patient will have 50mls of blood taken.Information about the patients ICU stay will also be recorded.

DETAILED DESCRIPTION:
Ceftolozane-tazobactam has recently emerged as a highly valuable option for the management of severe Gram-negative infections including those caused by multi-drug resistant (MDR) organisms, demonstrating superior antibacterial activity against the pathogens most frequently causing serious infection in the critically ill, such as Pseudomonas aeruginosa and Enterobacteriaceae spp, when compared with other commonly used beta-lactam antibiotics.

Although the continued reduction in the pathogen susceptibility to commonly used antibiotics in ICUs could be multifactorial, the potential contribution from inappropriate antibiotic exposure is undoubtedly very significant. Numerous clinical studies have reported sub-therapeutic antibiotic concentrations in ICU patients across different antibiotic classes, with conventional dosing regimens. This is due to marked changes in the pharmacokinetics (PK) and pharmacodynamics (PD) of antibiotics in the critically ill arising from disease-related physiological changes. Ceftolozane being a structural analogue of ceftazidime, shares similar PK properties of ceftazidime, and other beta-lactams, with a short half-life of about 2 hours, distribution into extracellular fluid, and predominant renal elimination, which all make it vulnerable to disease-related PK alterations in the critically ill.

Inappropriate antibiotic exposure in the ICU can also arise due to use of extracorporeal therapies such as continuous renal replacement therapy (CRRT). Many beta-lactam antibiotics share similar physicochemical and PK properties with ceftolozane and are efficiently cleared by CRRT machines. However the extent of total drug clearance during CRRT is variable not only due to the different modalities and operational settings across different institutions, but also due to the variable residual renal clearance associated with the degree of renal impairment. The traditional dosing considerations in patients undergoing CRRT mainly focus on the notion of renal impairment and generally consider low doses without giving appropriate consideration to the possibly high extracorporeal clearance, and thus risking under dosing. In a similar fashion, the product information for ceftolozane-tazobactam or the prescriber's information by the United States Food and Drug Administration (FDA), recommends a ten-fold lower-than-normal dose for use during renal replacement therapy (maintenance dose of 150mg versus 1.5g in those with normal renal function). However, to date there is limited data from clinical studies during CRRT in ICU patients to confirm if such a low dose provides appropriate antibiotic exposure. Lessons from studies on other beta-lactams suggest that ceftolozane may be subject to extensive but variable clearance during CRRT. It is therefore, essential to describe the adequacy of dosing in patients receiving CRRT, given that fact and that several additional pathophysiological factors affect the PK and PD of antibiotics even in the absence of extracorporeal circuits.

This prospective observational study will describe, firstly, the PK of ceftolozane-tazobactam in ICU patients who are not receiving CRRT, and secondly, the influence of CRRT on the PK and dosing requirements of ceftolozane-tazobactam in critically ill patients. This study will generate new PK data in ICU patients describing the exposure to ceftolozane-tazobactam from the recommended dosing regimen thereby allowing assessment of its adequacy and/or defining appropriate dosing. Further, it will provide invaluable insight into the altered dosing needs of patients receiving CRRT to enable its use in such patients through prediction of any necessary dosing corrections to account for the due effect of CRRT.

ELIGIBILITY:
Inclusion Criteria:

Group 1 Non CRRT

* Diagnosis of systemic infection known or suspected to be caused by an organism susceptible to ceftolozane-tazobactam
* Age more than 18 years
* The treating clinician considers Ceftolozane-tazobactam to be an appropriate agent to treat the infection Group 2 CRRT
* Diagnosis of systemic infection known or suspected to be caused by an organism susceptible to ceftolozane-tazobactam
* Age more than18 years
* Prescribed to receive CRRT
* The treating clinician considers Ceftolozane-tazobactam to be an appropriate agent to treat the infection

Exclusion Criteria:

Group 1 Non CRRT

* Renal dysfunction that necessitates the use of renal replacement therapy
* Known or suspected allergy to cephalosporins
* Receipt of any Pipercillin-Tazobactam for the treatment of this current infection.
* Pregnancy Group 2 CRRT
* Known or suspected allergy to cephalosporins
* Pregnancy
* Receipt of any Pipercillin-Tazobactam for the treatment of this current infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients receiving Ceftolozane-tazobactam for gram negative infection
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Roberts, Professor, Principal Investigator — Royal Brisbane and Womens Hospital
Locations (1):
- Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
All data will be reported and analysed in a de-identified format.

RESULTS

PARTICIPANT FLOW:
Groups:
- CRRT Group: Critically ill patients receiving Ceftolozane-Tazobactam who require continuous renal replacement therapy
  CRRT group: CRRT group: Pre and Post dialysis filter blood samples taken prior to first dose of Ceftolozane-tazobactam and at 15min, 45min, 1h 2h 3h 4h 5h 6h 7h 8h.
  Ultrafiltrate samples at 1 hr,2h 4h 6h 8h
Period: Overall Study
Arm/Group | Non CRRT Group | CRRT Group
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non CRRT Group | CRRT Group | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 56 [52 to 61] | 61.5 [58 to 65] | 58 [51.5 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Serum Creatinine [Median (Inter-Quartile Range); unit: micro-mole/litre] | 46 [39 to 77] | 138 [92 to 151.75] | 75 [42.5 to 138]

OUTCOME MEASURES:

1. Primary Outcome: Probability of Target Attainment for 40% fT>MIC
Description: The probability of attaining free concentrations above MIC for 40% of the time
Time Frame: 24 hour period
Population: For a recommended dose of 1.5g every 8 hours for patients without CRRT and for a dosing regimen of 3g loading dose plus 0.75 g every 8 hours for patients with CRRT when evaluated at the EUCAST MIC breakpoint of 4mg/L for Pseudomonas aeruginosa
Measure: Number; unit: percentage of time above MIC
Arm/Group | Non CRRT Group | CRRT Group
Number analyzed (Participants) | 12 | 6
percentage of time above MIC | 100 | 100

ADVERSE EVENTS:
Time Frame: 1week
Description: This study was observational pharmacokinetic study and not an outcomes study. No drug-related adverse events were observed during the study sampling period.
  "0" Total Number of Participants at Risk means that "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Non CRRT Group | CRRT Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT02962934/Prot_SAP_000.pdf